CLINICAL TRIAL: NCT00708617
Title: Non Invasive Diagnostic Methods for Fibrosis in Alcoholic Liver Disease : FIBROSCAN Validation and Comparison of Fibrotest - FIBROSCAN Association With FIBROSCAN Alone
Brief Title: FIBROSCAN Validation and Interest of Fibrotest - FIBROSCAN Association for Fibrosis Diagnosis in Alcoholic Liver Disease
Acronym: FIBROMAF
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Echosens (Industry)
Responsible Party: Sponsor
Other Study IDs: OST07008
Record Dates: First submitted 2008-07-01; First posted 2008-07-02 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Alcoholic Liver Disease
Keywords: Liver fibrosis; Alcoholic liver disease; Non invasive diagnostic methods; Transient elastography; Fibrotest
MeSH Terms: conditions — Liver Diseases, Alcoholic; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Apart from Fibrotest, non-invasive markers have been validated only for chronic hepatitis C. However as for chronic C hepatitis, non invasive tests (Fibrotest and transient elastometry) are already used in current practice. The aim of this study is to validate the diagnostic value of FIBROSCAN by comparison with liver histology. FIBROSCAN will be also compared to Fibrotest and FIBROSCAN-Fibrotest association to each test alone in order to optimize this diagnostic strategy.

Studied variables will be significant fibrosis (≥ 2 in the METAVIR score) and presence of cirrhosis (score : F4). Diagnostic values of the scores will be expressed by sensitivity, specificity, positive and negative predictive values, and ROC curves. Areas under ROC curve of the scores will be compared using Z test.

DETAILED DESCRIPTION:
Alcoholic liver disease (ALD) is highly prevalent and liver fibrosis and cirrhosis are asymptomatic for a long time. Liver biopsy in patients with ALD is designed to determine the prognostic of the liver lesions and to manage cirrhosis. Apart from Fibrotest, non-invasive markers have been validated only for chronic hepatitis C. However as for chronic C hepatitis, non invasive tests (Fibrotest and transient elastometry) are already used in current practice. The aim of this study is to validate the diagnostic value of FIBROSCAN by comparison with liver histology. FIBROSCAN will be also compared to Fibrotest and FIBROSCAN-Fibrotest association to each test alone in order to optimize this diagnostic strategy.

200 consecutive excessive drinkers with aminotransferase anomalies or suspicion of cirrhosis will be included in the study over a period of 2 years. All patient will have intercostal liver biopsy, assessment of the non-invasive biological scores of liver fibrosis and transient elastography.

Studied variables will be significant fibrosis (≥ 2 in the METAVIR score) and presence of cirrhosis (score : F4). Diagnostic values of the scores will be expressed by sensitivity, specificity, positive and negative predictive values, and ROC curves. Areas under ROC curve of the scores will be compared using Z test. Multivariate analyses will be used to identify the scores with an independent diagnostic value and therefore that could be associated.

This study will allow to select the non-invasive marker(s) with the best diagnostic values in order to identify early fibrosis in patients with ALD.

ELIGIBILITY:
Inclusion Criteria:

* consecutive excessive drinkers
* both gender
* aged 18 to 75 years,
* hospitalized to manage alcoholic liver disease
* Ag HBs -, HIV -, HCV -, without any other liver disease than alcohol abuse,
* with alcohol consumption greater than 80 g per day for at least 5 years
* with aminotransferase levels anomalies (ASAT ≥ 1.5 N and ALAT > N) or suspicion of cirrhosis

Exclusion Criteria:

* any other liver disease than alcohol abuse,
* ascitis,
* contraindication to intercostal liver biopsy
* IMC>30
* liver carcinoma
* other carcinoma
* serious associate disease
* platelets < 60 GIGAS/L or Quick time < 50% or TCA > 1.5 witness time
* treatment with Plavix® or platelet antiaggregant or anticoagulant
* intercostal liver biopsy refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alcoholic Liver Disease
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2008-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Patients will be classified according to existence of significant fibrosis (METAVIR score>=2)and cirrhosis (METAVIR score=4) Areas under ROC curve of the diagnostic tests | up to one week

SECONDARY OUTCOMES:
Diagnostic values of the diagnostic tests will be expressed by sensitivity, specificity, positive and negative predictive values, and ROC curves. | up to one week

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Naveau, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris Hôpital Antoine Béclère
Locations (3):
- France (3):
  - AP-HP Hôpital Antoine Beclere, Clamart
  - Hôpital Claude Huriez, Lille
  - AP-HP Hôpital Cochin, Paris